CLINICAL TRIAL: NCT00522561
Title: Lower Limb Mechanical Characteristics: Effect on Running Mechanics and Energetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Roger Oullion, Centre Hospitalier Universitaire de Saint-Etienne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0701039; 2007-A00562-51; DGS 2007-0360
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Healthy volunteers; running; energetic cost; limb mechanical characteristics; contractile components; elastic components; healthy men doing regularly physical activities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): healthy volunteers
  Interventions: Other: energetic and non invasive limb mechanical measurements

INTERVENTIONS:
Other: energetic and non invasive limb mechanical measurements — Force velocity stiffness running

SUMMARY:
Inter-individual variability in energetic cost of running may be partly explained by lower limbs mechanical characteristics. The transposition of muscle mechanical model with two components (contractile and elastic) to the whole lower limb mechanical behavior analysis during running. The main aim of present investigation is to study the effects of lower limb mechanical characteristic (force, velocity, stiffness) on the energetic cost of running using a lower limb mechanical approach including both contractile and elastic components.Twenty healthy men will run on a treadmill at 12km.h-1 in 8 different 5 min-conditions. Through conditions, stride frequency, sole stiffness and subject's body weight will be changed to allow artificial variations in lower limb mechanical characteristics. Energetic and non-invasive mechanical measurements analysis will be performed to obtain energetic cost of running and to compute force, velocity and stiffness of lower limbs for each condition.

DETAILED DESCRIPTION:
Main aim: Identify the effect of mechanical characteristic induced on lower limbs on the energetic cost of running.

Secondary aim : Minimize the energetic cost of running by lower limb mechanical characteristics optimization.

ELIGIBILITY:
Inclusion Criteria:

* healthy men being between 20 and 35 years old and doing regularly physical activities
* subjects must be able to run at 12 km/h during 15 minutes in aerobic condition
* not be sedentary and not do running competitions
* be affiliated to a social security system
* Sign a written inform consent

Exclusion Criteria:

* presenting a clinic sign of intolerance to exercise, and particularly to running
* overweight subjects
* having a medical treatment which may interfere with the running quality or with one of the physiological parameters measured
* taking part at the same moment in another medicinal research

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
the energetic cost of running: the energetic cost (Oxygen consumption by meter covered) is calculated by the ratio of oxygen consumption on the running velocity. | within 4 weeks after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Roger OULLION, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Service de Physiologie clinique et de l'exercice - CHU Saint-Etienne, Saint-Etienne, France